CLINICAL TRIAL: NCT03076658
Title: Open Access Database of Standing Full Body Radiographs in Asymptomatic Volunteers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15-2433
Record Dates: First submitted 2017-01-11; First posted 2017-03-10 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Intervertebral Disc Degeneration; Osteoarthritis, Spine
MeSH Terms: conditions — Intervertebral Disc Degeneration; Osteoarthritis, Spine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- asymptomatic EOS Imaging (Other): patients that qualify for study and EOS imaging to analyze spino-pelvic parameters
  Interventions: Radiation: EOS imaging

INTERVENTIONS:
Radiation: EOS imaging — The EOS imaging system will be utilized to obtain full-body radiographs in frontal and sagittal projections obtained in the upright standing position. Measurements will include a coronal plumb-line, sagittal vertebral axis (SVA), external auditory meatus plumb-line, cervical lordosis, thoracic kyphosis, lumbar lordosis, hip flexion/extension, knee flexion/extension, ankle flexion/extension, T1 tilt, T1 spino-pelvic instance, acetabular index, pelvic tilt (PT), pelvic incidence (PI), and sacral slope (SS).

SUMMARY:
A study of the skeletal structure and how the structure changes over time. The aim of the study is to evaluate the skeleton in 10 year increments to determine an understanding of the normal skeleton as a person ages. By using x-ray analysis, a new low dose x-ray system (EOS) can be used to evaluate the whole body to see changes in the bone structure over time. Subjects will be asked to undertake one x-ray analysis of their whole body skeletal structure. There will be 25 male and 25 female subjects per decade. The averaging of the measured skeletal parameters will provide information on changes over time generating a standardized expectation of general changes in skeletal structure as participants age.

DETAILED DESCRIPTION:
Current techniques of advanced spinal surgery allow physicians to correct complex spinal deformity to nearly any alignment desired. The investigators ability to analyze spino-pelvic alignment has evolved concurrently; however, the investigators goals in deformity correction are still not completely understood. With increasing ability to assess whole body alignment, the investigators must establish a baseline for the "normal" population inclusive of age related changes. the investigators hypothesis is that global body alignment will vary based on sex and progressively vary with age.

The goal of this study is to create an open access database of "normal" volunteer full body radiographic images obtained using the new EOS biplanar x-ray imaging system. The system provides a radiographic view of the weight-bearing skeleton equivalent to plain radiography. The development of an open access database of full body images and global spine parameters will provide spine surgeons with normative data that can be used to guide clinical decision making and surgical planning. Furthermore, the database can be used by researchers to obtain control measurements for comparison in studies of various spine, and potentially non-spine, pathologies.

Specific Aims

1. To create an open access database of radiographic full body images in the sagittal and coronal planes of subjectswithout spine deformities or acute or severe chronic disease, across a range of age groups from 20 to 80 year old males and females.
2. To document age related changes that occur in radiographic parameters in the spine and pelvis by including subjects across a wide range of ages.

ELIGIBILITY:
Inclusion Criteria:

* Males and females age 21-85 without a history of spine surgery.

Exclusion Criteria:

* History of spine or neural axis surgery
* History of cancer with or without metastatic disease
* Connective tissue, rheumatologic (or other inflammatory arthropathies), or neurologic disorders
* History of knee replacement surgery, as these may have contractures causing unexpected changes in alignment
* Severe osteoarthritis of the hips/knees/ankles
* Spondylitis
* Compression fractures or other trauma of the spinal column
* Previous trauma/fractures of the pelvis whether or not surgery was required
* Previous trauma or fractures of the lower extremities requiring surgery
* Pregnant women
* BMI >37
* Oswestry Disability Index score >25

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-09; Primary Completion 2031-01 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Coronal plumb-line | Through 1 EOS scan, 20 minutes
Sagittal vertebral axis (SVA) | Through 1 EOS scan, 20 minutes
External auditory meatus plumb-line | Through 1 EOS scan, 20 minutes
Cervical lordosis | Through 1 EOS scan, 20 minutes
Thoracic kyphosis | Through 1 EOS scan, 20 minutes
Lumbar lordosis | Through 1 EOS scan, 20 minutes
Hip flexion/extension | Through 1 EOS scan, 20 minutes
Knee flexion/extension | Through 1 EOS scan, 20 minutes
Ankle flexion/extension | Through 1 EOS scan, 20 minutes
T1 tilt | Through 1 EOS scan, 20 minutes
T1 spino-pelvic instance | Through 1 EOS scan, 20 minutes
Acetabular index | Through 1 EOS scan, 20 minutes
Pelvic tilt (PT) | Through 1 EOS scan, 20 minutes
Pelvic incidence (PI) | Through 1 EOS scan, 20 minutes
Sacral slope (SS) | Through 1 EOS scan, 20 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Kleck, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Coloardo Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Researchers, at the end of the study, can make data request to Principle Investigator and then requested data can be obtained via RedCap.